CLINICAL TRIAL: NCT00357981
Title: Patient Experiences Using Evra for Management of Menstrual Related Symptoms.
Brief Title: Continuous Use of the Contraceptive Patch and the Personal Economic Impact.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Both sponsor and UCSF decided this study was not clinical relevant at this time
Sponsor: University of California, San Francisco (Other)
Collaborators: Ortho-McNeil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10857-25721-01
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Dysmenorrhea; Menstruation Disturbances; Menstruation Disorders
Keywords: Contraceptive patch; menstruation; economics
MeSH Terms: conditions — Dysmenorrhea; Menstruation Disturbances | interventions — Ortho Evra

ARMS (1):
- ORTHO EVRA (Experimental): The approximate first two months of women's participation will be spent documenting baseline information about their health and well-being, work patterns and performance, and the economic impact of their menstruation. Subjects will then initiate two, two month intervals of continuous use of ORTHO EVRA.
  Over this four month treatment period, subjects will document their health and well-being, work patterns and performance, and the economic impact of their menstruation while being treated with ORTHO EVRA. This will allow us to compare subjects' experiences pre- and post-treatment. The study's instruments will focus on eliciting information on the personal and economic costs of menstruation such as measuring time missed from work, changes in productivity and work satisfaction, and impact on quality of life.
  Interventions: Drug: ORTHO EVRA, the contraceptive patch

INTERVENTIONS:
Drug: ORTHO EVRA, the contraceptive patch

SUMMARY:
Dr. Eleanor Drey in the Department of Obstetrics, Gynecology and Reproductive Sciences UCSF is conducting a study to examine the personal and economic impact of continuous use of ORTHO EVRA, the contraceptive patch, on menstrual related symptoms for women who report having severe menstrual related symptoms.

DETAILED DESCRIPTION:
30 adult women, 18-40 years of age, will be recruited to participate in a six month study. The focus of recruitment will be on women with menstrual-related symptoms who are currently working in physically demanding, low autonomous service jobs.

The approximate first two months of women's participation will be spent documenting baseline information about their health and well-being, work patterns and performance, and the economic impact of their menstruation. Subjects will then initiate two, two month intervals of continuous use of ORTHO EVRA.

Over this four month treatment period, subjects will document their health and well-being, work patterns and performance, and the economic impact of their menstruation while being treated with ORTHO EVRA. This will allow us to compare subjects' experiences pre- and post-treatment. The study's instruments will focus on eliciting information on the personal and economic costs of menstruation such as measuring time missed from work, changes in productivity and work satisfaction, and impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, women 18 through 40 years of age at the time of enrollment who have severe menstrual related symptoms
* Willing and able to comply with the study protocol
* Has not used oral contraceptives, vaginal rings, or injectable contraceptives during the last month and has had one regular menstrual period preceding enrollment OR is within seven days post induced abortion
* Has been determined to be eligible for hormonal contraceptive use
* Willing and able to be contacted by research staff.

Exclusion Criteria:

* Does not speak or read English
* Is breastfeeding
* Has contraindications to use of estrogen-containing contraceptives including thrombophlebitis or thromboembolic disorders including a past history of deep vein thrombophlebitis or thromboembolic disorders
* Cerebrovascular or coronary artery disease
* Known or suspected carcinoma of the breast, endometrium or suspected estrogen-dependent neoplasia
* Undiagnosed abnormal genital bleeding
* Biliary tract disease
* Cholestatic jaundice of pregnancy or jaundice with prior contraceptive steroid use
* Hepatitis
* Cirrhosis
* Hepatic adenomas or carcinoma
* Hypertension (>140 systolic or >90 diastolic)
* Diabetes
* Migraine with focal neurologic symptoms
* Is pregnant or less than 3 months postpartum
* Concurrent use of medications that induce liver enzymes
* Has severe or chronic constipation
* Drug or alcohol abuse (current or within the last 12 months)
* Unable or unwilling to comply with protocol
* Is HIV-positive
* Has history or presence of cancer
* Treatment (other than hormonal contraception) has been recommended for menstrual symptoms
* Taking prescription medication because of menstrual related symptoms

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Birth control satisfaction after four months of patch use | Four months
Health-related work productivity scales after four months of patch use | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Drey, MD, EdM, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Background] Cote I, Jacobs P, Cumming D. Work loss associated with increased menstrual loss in the United States. Obstet Gynecol. 2002 Oct;100(4):683-7. doi: 10.1016/s0029-7844(02)02094-x. PMID 12383534
- [Background] Dawood MY. Nonsteroidal anti-inflammatory drugs and changing attitudes toward dysmenorrhea. Am J Med. 1988 May 20;84(5A):23-9. doi: 10.1016/0002-9343(88)90473-1. PMID 3287908
- [Background] Kristjansdottir J, Johansson ED, Ruusuvaara L. The cost of the menstrual cycle in young Swedish women. Eur J Contracept Reprod Health Care. 2000 Jun;5(2):152-6. doi: 10.1080/13625180008500385. PMID 10943579
- [Background] Braunstein JB, Hausfeld J, Hausfeld J, London A. Economics of reducing menstruation with trimonthly-cycle oral contraceptive therapy: comparison with standard-cycle regimens. Obstet Gynecol. 2003 Oct;102(4):699-708. doi: 10.1016/s0029-7844(03)00738-5. PMID 14550999
- [Background] Kjerulff KH, Erickson BA, Langenberg PW. Chronic gynecological conditions reported by US women: findings from the National Health Interview Survey, 1984 to 1992. Am J Public Health. 1996 Feb;86(2):195-9. doi: 10.2105/ajph.86.2.195. PMID 8633735
- [Background] Kaunitz AM. Menstruation: choosing whether...and when. Contraception. 2000 Dec;62(6):277-84. doi: 10.1016/s0010-7824(00)00182-7. PMID 11239613